CLINICAL TRIAL: NCT05704400
Title: Efficacy of Chimeric Monoclonal Anti-CD20 Antibodies (Rituximab Biosimilar) Associated With Monoclonal Anti-CD38 (Daratumumab) in the Treatment of Childhood Multidrug Dependent and Resistant (MDNS, MRNS) Nephrotic Syndrome
Brief Title: Efficacy of Anti-CD20 Ab Associated With Anti-CD38 in the Childhood Multidrug Dependent and Resistant Nephrotic Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Giannina Gaslini (Other)
Responsible Party: Principal Investigator, Gian Marco Ghiggeri MD, PhD, Principal Investigator, Istituto Giannina Gaslini
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DUAL1
Record Dates: First submitted 2022-12-16; First posted 2023-01-30 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Nephrotic Syndrome
MeSH Terms: conditions — Nephrotic Syndrome | interventions — daratumumab

STUDY DESIGN:
Intervention Model Description: Phase II Proof of concept, the Dual 1 is a before-after clinical trial testing the superiority of rituximab plus daratumumab in maintaining drug free disease remission in patients with multi-drug dependent nephrotic syndrome
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- single arm (Experimental)
  Interventions: Drug: Rituximab Biosimilar ABP 798; Drug: Daratumumab

INTERVENTIONS:
Drug: Rituximab Biosimilar ABP 798 — Rituximab IV: the dose is standard for pediatric nephrotic syndrome; for dosage between 100 and 250 mg rituximab will be diluted in 100 ml of normal saline and administered at 2 ml/h for the first 30'; 3 ml/h for the second 30'; 6 ml/h for the third 30'; 15 ml/h until the end. For dosage between 260 and 500 mg rituximab will be diluted in 250 ml of normal saline and administered at 6 ml/h for the first 30'; 9 ml/h for the second 30'; 18 ml/h for the third 30'; 36 ml/h until the end. For dosage between 510 and 1000 mg rituximab will be diluted in 500 ml of normal saline and administered at 9 ml/h for the first 30'; thereafter, the infusion rate can be doubled every 30 minutes up to a maximum of 72 ml/h.
Drug: Daratumumab — Daratumumab vials 20 mg 1 ml will be collected to reach the desired dose of 16 mg /Kg, the dose is standard recommend to treat myeloma; diluted in 1000 ml of normal saline and infused at the constant speed of 50 ml/h. This will be reduced in case of cutaneous allergic reactions

SUMMARY:
Nephrotic syndrome is considered a disease caused by an interplay of immunological stimuli with adaptive immunity(CD80/CD40) as trigger and Treg in the mid between co-stimulatory molecules and effectors. The positive effect of drugs blocking CD20 maturation in SDNS suggests a main role of these cells in regulating the system. Multidrug dependent, multidrug resistant nephrotic syndrome as well as post transplant FSGS recurrence patients can be considered difficult to treat patients and the association of two drugs, one targeting CD20 and a targeting plasmacells can be use in order to block the stimulatory cascade at more sites.

DETAILED DESCRIPTION:
Nephrotic syndrome is considered a disease caused by an interplay of immunological stimuli with adaptive immunity(CD80/CD40) as trigger and Treg in the mid between co-stimulatory molecules and effectors. The positive effect of drugs blocking CD20 maturation in SDNS suggests a main role of these cells in regulating the system. One possible explanation of proteinuria resolution by anti-CD 20 in most but not all patients with SDNS/MDNS is that some CD20 cells may escape the inhibition and mature in some cases to plasmacells. On this basis, it seems reasonable to consider the association of two drugs, one targeting CD20 and one targeting plasmacells in order to block the stimulatory cascade at more sites. There are recent positive evidences from the association of 2 monoclonal antibodies that block maturation of CD20 at different steps. One study utilized the humanized anti-CD20 antibody obinutuzumab(single dose 1,000 mg 1.73m2) in combination with the anti-CD38 (plasmacells) monoclonal antibody daratumumab (1,000 mg 1.73m2)18 in patients who relapsed after conventional treatments with Prednisone, rituximab and CNI and developed dependence to the combination of more than 2 drugs (MDNS). A cohort of 14 patients treated with the above association were included in a retrospective analysis: all of them suspended oral drugs, 5 out of 14 presented recurrence of proteinuria after about 10 months, 9 out of 14 were in stable remission after 20 months. Therefore, the use of 2 monoclonal antibodies in low doses is potentially valuable considering the positive results and also taking in account the safety of the treatment. While it is not possible to discern the separate effects of obinutuzumab and daratumumab when given together, the preliminary positive results of their combination may open new ways in the treatment of nephrotic syndrome and supports the necessity of new studies in those patients who require more than one drug to maintain remission. The investigators hypothesize that rituximab in place of obinutuzumab (not available in Italy for the use in nephrotic syndrome) with daratumumab could produce the same positive effects in MDNS and MRNS.

The Dual 1 is a before-after clinical trial testing the superiority of rituximab plus daratumumab in maintaining drug free disease remission in patients with multi-drug dependent nephrotic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age between 3 and 24 years
* Multidrug dependent or resistant nephrotic syndrome for at least six months before enrolment. The need of at least 2 of the oral drugs listed below defines multidrug-dependence: prednisone at any doses, MMF 1200 mg m2 and CNI 0.1 mg day given in two doses. Dependence is defined by two consecutive relapses during double therapies or within 14 days of ceasing one of the three components of the therapeutic approach. Resistance is defined as lack of antiproteinuric effect of a double therapy based on steroid plusCNI or mofetilmycophenolate (MMF).Steroid resistance is defined by failure to achieve complete remission after 6 weeks with prednisone60 mg/m2.
* Post transplant recurrence of FSGS.
* Ability to provide consent and assent: parents'/guardian's written informed consent, and child's assent given before any study-related procedure not part of the subject's normal medical care, with the understanding that consent may be withdrawn by the subject any time without prejudice to his or her future medical care.

Exclusion Criteria:

* Positivity to autoimmunity tests (ANA, nDNA, ANCA)
* Reduction of C3 levels.
* eGFR<60/ml/min/1,73 m2 valuated according to revised Bedside Schwartz Formula for patients between 2 and 17 years and with CKD-EPI Creatinine 2009 Equation for 18 years old patients.
* Pregnancy
* Neoplasm
* Infections: previous or actual HBV (with HBeAb positivity) or HCV infection
* CD20 B lymphocytes count <2,5%
* Treatment with Rituximab or cyclophosphamide in the last 6 months

Ages: 3 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Safety- number of treatment-related adverse events | 12 months
  Primary: to test whether the combination of rituximab and daratumumab is safe and can achieve and maintain drug-free disease remission in patients with multi drug-dependent nephrotic syndrome within 12 months. The investigators will consider the number of participants with treatment-related adverse events as assessed by CTCAE v4.0 This outcome will not be compared but only studied following the intervention.
Efficacy- number of months in remission | 12 months
  To test whether the combination of rituximab and daratumumab can achieve and maintain drug-free disease remission in patients with multi drug-dependent nephrotic syndrome within 12 months The investigators will compare the outcome of log-albuminuria following the infusion of the two drugs to the log-albuminuria before the infusion, when patients were maintained by the association of MMF and CNI (i.e. the drug recommended by Clinical Practice Guidelines-KDIGO as benchmark of the treatment).

SECONDARY OUTCOMES:
Prediction | 12 months
  To analyze B and T cell lymphocyte subsets pre and post-therapy with Rituximab/Daratumumab

CONTACTS AND LOCATIONS:
Overall Officials: Gianmarco Ghiggeri, MD, Principal Investigator — IRCCS G. Gaslini
Locations (1):
- IRCCS G. Gaslini, Genova, Italy

IPD SHARING:
Plan to Share IPD: Yes
The completed study will be summarized in a final report that accurately and completely presents the study objectives, methods, results, limitations of the study, and interpretation of findings.
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Derived] Angeletti A, Bruschi M, Kajana X, La Porta E, Spinelli S, Caridi G, Lugani F, Verrina EE, Ghiggeri GM. Biologics in steroid resistant nephrotic syndrome in childhood: review and new hypothesis-driven treatment. Front Immunol. 2023 Aug 29;14:1213203. doi: 10.3389/fimmu.2023.1213203. eCollection 2023. PMID 37705972